CLINICAL TRIAL: NCT02122341
Title: Post FDA-Approval Clinical Evaluation of BackStopTM in Patients Undergoing Ureteroscopic Lithotripsy: A Prospective, Randomized Clinical Trial
Brief Title: Clinical Evaluation of BackStop in Patients Undergoing Ureteroscopic Lithotripsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has halted prematurely as we were not able to meet our target accrual.
Sponsor: University of Southern California (Other)
Collaborators: Urology of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-12-00714
Record Dates: First submitted 2014-04-18; First posted 2014-04-24 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BackStop (Experimental): Patients randomized to the Experimental arm will receive the BackStop gel during their ureteroscopic lithotripsy to prevent retrograde migration of stones or stone fragments.
  Interventions: Device: BackStop
- Control (No Intervention): Patients randomized to the control group will not use any devices to prevent retrograde migration of stones and stone fragments during their ureteroscopic lithotripsy.

INTERVENTIONS:
Device: BackStop — BackStop™ is a FDA approved device. It is intended for use during ureteroscopic lithotripsy to prevent retrograde migration of stones and stone fragments. It is comprised of a solution of a thermosensitive polymer, a purified version of poloxamer 407 having been fractionated in saline. BackStop™, which is injected above the stone, is provided in sterile, pre-filled 2.5ml and 5ml syringes along with and a corresponding injector and a catheter (3F or 5F).
  Arms: BackStop

SUMMARY:
The purpose of this clinical study is to evaluate BackStop, a polymer-based device that is intended to be used during ureteroscopic lithotripsy to prevent retrograde stone migration.

DETAILED DESCRIPTION:
During ureteroscopic treatment for ureteral stones, lithotripsy, irrigation, and manipulation of the stone often pushes stone away into the kidney itself. This phenomenon is called retropulsion, which is defined as clinically significant retrograde migration of stone or stone fragments. Movement of stones retrograde into the renal pelvis could potentially add and complicate the surgery further. Often scopes need to be changed in order to reach the stone, and chasing these stones will add time to the surgery and require more valuable resources. Furthermore, sometimes a second operation will need to be done when these retropulsed fragments could not be all found and cleaned out.

A number of devices have been developed to prevent such migration including stone baskets and conical devices. These are wire-based devices which have the potential of injuring the ureter. Because of safety concerns and that there is limited data available on the effectiveness of these devices; these are not widely used by urologists. BackStop has recently been developed as another tool to prevent retropulsion. It is a water soluble gel that is injected proximal to the stone. This creates a physical barrier that prevents stone migration during ureteroscopic lithotripsy for ureteral calculus.

ELIGIBILITY:
Inclusion Criteria:

* patient with solitary ureteral stone ranging from 5mm to 15mm diameter
* able to tolerate general anesthesia
* clinical indication for treatment by ureteroscopic lithotripsy
* must be willing and able to participate in any follow-up visits
* provide informed consent
* have a CT scan demonstrating the stone

Exclusion Criteria:

* patients undergoing extracorporeal shock wave lithotripsy (ESWL) or any other extracorporeal or percutaneous lithotripsy procedure as primary procedure
* any co-morbidity or condition that would necessitate exclusion of patient (physician opinion)
* renal or ureteral anatomical abnormality
* multiple stones in the indicated ureter
* stones in the indicated kidney
* patient is immunocompromised
* multiple organ dysfunction syndrome
* has an absolute or relative solitary kidney mass
* >= Stage 3 chronic kidney disease
* bilateral ureteral obstructing stones
* staghorn calculi
* impaction of several stone fragments (Steinstrasse)
* uncorrected coagulopathy/thrombocytopenia
* urethral and/or ureteral stricture
* reconstructive urinary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Dunn, M.D., Principal Investigator — USC Institute of Urology
Locations (2):
- United States (2):
  - USC Institute of Urology, Los Angeles, California
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segura JW, Preminger GM, Assimos DG, Dretler SP, Kahn RI, Lingeman JE, Macaluso JN Jr. Ureteral Stones Clinical Guidelines Panel summary report on the management of ureteral calculi. The American Urological Association. J Urol. 1997 Nov;158(5):1915-21. doi: 10.1016/s0022-5347(01)64173-9. PMID 9334635
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Background] Hendrikx AJ, Strijbos WE, de Knijff DW, Kums JJ, Doesburg WH, Lemmens WA. Treatment for extended-mid and distal ureteral stones: SWL or ureteroscopy? Results of a multicenter study. J Endourol. 1999 Dec;13(10):727-33. doi: 10.1089/end.1999.13.727. PMID 10646679
- [Background] Pardalidis NP, Kosmaoglou EV, Kapotis CG. Endoscopy vs. extracorporeal shockwave lithotripsy in the treatment of distal ureteral stones: ten years' experience. J Endourol. 1999 Apr;13(3):161-4. doi: 10.1089/end.1999.13.161. PMID 10360494
- [Background] Chow GK, Patterson DE, Blute ML, Segura JW. Ureteroscopy: effect of technology and technique on clinical practice. J Urol. 2003 Jul;170(1):99-102. doi: 10.1097/01.ju.0000070883.44091.24. PMID 12796655
- [Background] Knispel HH, Klan R, Heicappell R, Miller K. Pneumatic lithotripsy applied through deflected working channel of miniureteroscope: results in 143 patients. J Endourol. 1998 Dec;12(6):513-5. doi: 10.1089/end.1998.12.513. PMID 9895254
- [Background] Robert M, Bennani A, Guiter J, Averous M, Grasset D. Treatment of 150 ureteric calculi with the Lithoclast. Eur Urol. 1994;26(3):212-5. doi: 10.1159/000475382. PMID 7805707
- [Background] Rane A, Bradoo A, Rao P, Shivde S, Elhilali M, Anidjar M, Pace K, D'A Honey JR. The use of a novel reverse thermosensitive polymer to prevent ureteral stone retropulsion during intracorporeal lithotripsy: a randomized, controlled trial. J Urol. 2010 Apr;183(4):1417-21. doi: 10.1016/j.juro.2009.12.023. Epub 2010 Feb 20. PMID 20171695
- See also: FDA MAUDE database online (accessed date July 8, 2007) — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfMAUDE/TextSearch.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: BackStop: Patients randomized to the Experimental arm will receive the BackStop gel during their ureteroscopic lithotripsy to prevent retrograde migration of stones or stone fragments.
  BackStop: BackStop™ is a FDA approved device. It is intended for use during ureteroscopic lithotripsy to prevent retrograde migration of stones and stone fragments. It is comprised of a solution of a thermosensitive polymer, a purified version of poloxamer 407 having been fractionated in saline. BackStop™, which is injected above the stone, is provided in sterile, pre-filled 2.5ml and 5ml syringes along with and a corresponding injector and a catheter (3F or 5F).
- No Intervention: Control: Patients randomized to the control group will not use any devices to prevent retrograde migration of stones and stone fragments during their ureteroscopic lithotripsy.
Period: Overall Study
Arm/Group | Experimental: BackStop | No Intervention: Control
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Backstop | No Intervention: Control | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 13 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Rate of Prevention of Retrograde Stone or Stone Fragment Migration
Description: Prevention of retrograde stone migration (Yes/No)
Time Frame: At the time of surgery
Measure: Count of Participants; unit: Participants
Groups:
- Investigational: BackStop: Patients randomized to the Experimental arm will receive the BackStop gel during their ureteroscopic lithotripsy to prevent retrograde migration of stones or stone fragments.
  BackStop: BackStop™ is a FDA approved device. It is intended for use during ureteroscopic lithotripsy to prevent retrograde migration of stones and stone fragments. It is comprised of a solution of a thermosensitive polymer, a purified version of poloxamer 407 having been fractionated in saline. BackStop™, which is injected above the stone, is provided in sterile, pre-filled 2.5ml and 5ml syringes along with and a corresponding injector and a catheter (3F or 5F).
Arm/Group | Investigational: BackStop | No Intervention: Control
Number analyzed (Participants) | 17 | 18
Participants
  Yes | 14 | 11
  No | 3 | 7

2. Secondary Outcome: Stone-free Rate
Description: Presence or absence of residual stone fragments at 2 month follow up after lithotripsy
Time Frame: 2 months
Population: Number of patients analyzed is inconsistent with numbers provided in participant flow module due to patients lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational: BackStop | No Intervention: Control
Number analyzed (Participants) | 9 | 10
Participants
  Present | 9 | 10
  Absent | 0 | 0

3. Other Pre Specified Outcome: Need for Secondary Procedures
Description: Need for secondary procedures of patients who had stone migration
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational: BackStop | No Intervention: Control
Number analyzed (Participants) | 3 | 7
Participants
  Yes | 0 | 0
  No | 3 | 7

4. Other Pre Specified Outcome: Time for BackStop Injection
Description: Time required to deliver BackStop beginning with insertion of BackStop catheter and ending with its removal subsequent to the delivery of BackStop
Time Frame: Minutes during Surgery
Population: The control group did not receive BackStop injection
Measure: Mean (Full Range); unit: minutes
Arm/Group | Investigational: BackStop | No Intervention: Control
Number analyzed (Participants) | 17 | 0
minutes | 3.04 [.43 to 14] |

5. Other Pre Specified Outcome: Duration of Lithotripsy Procedure
Description: Duration of Lithotripsy Procedure
Time Frame: during surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Investigational: BackStop | No Intervention: Control
Number analyzed (Participants) | 17 | 18
minutes | 4.17 [.08 to 30] | 6.09 [.1 to 28]

ADVERSE EVENTS:
Arm/Group | Investigational: BackStop | No Intervention: Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 4/17 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational: BackStop (N=17) | No Intervention: Control (N=18)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — Total of 3 participants experienced an adverse event that was not unexpected for standard lithotripsy procedure. None were attributed to BackStop.
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
Urethral Pain (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was not able to meet target accrual and was closed early. More patients are needed to fully evaluate the clinical effectiveness of BackStop.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No